CLINICAL TRIAL: NCT06398093
Title: Developing and Testing a Self-Compassion Tool Kit to Improve the Care of Individuals With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Chao, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 810394
Record Dates: First submitted 2024-04-28; First posted 2024-05-03 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Compassion Toolkit (Experimental)
  Interventions: Behavioral: Self-Compassion Tool Kit

INTERVENTIONS:
Behavioral: Self-Compassion Tool Kit — Participants will mediate, journal their reactions, exercise, and apply sleep hygiene measures over the course of four weeks.

SUMMARY:
There is a high prevalence of anxiety and depression in patients with Type 2 Diabetes (T2D). While past studies demonstrate the potential therapeutic effect of mindfulness-based interventions in patients with T2D, little is understood about the mode of delivery or quantity of the intervention necessary to experience benefits. This project aims to develop and implement a self-compassion tool kit based on the principles of mindfulness and meditation to better understand how self-compassion works to affect psychological health and wellbeing in patients with T2D. The investigators will study the impact of a self-compassion tool kit - including mindfulness meditation, exercise, journaling and sleep parameters - on T2D. Enhancing emotional well-being could complement current T2D treatments to facilitate improved quality of life.

DETAILED DESCRIPTION:
A pre-test and post-test experimental design will be used to evaluate the efficacy of the self-compassion tool kit on distress, coping, testing glucose, sleep, and wellness in adults living with T2D.

For this 4-week study, participants will receive education on Sleep Hygiene practices during the first week of the intervention. Mindfulness meditation will be offered to participants using the Headspace app and four, ten-minute sessions will be prescribed per week. For exercise, 30-60 minutes of daily physical activity will be prescribed and participants can select the exercise of their choice. Additionally, participants will receive a journal in the mail with prompts associated with each day of required journalling. Prompts will elicit reflections, gratitude and growth. Participants will be followed by telephone every week. Baseline and week four data will be collected using the Demographic Form, T2DDAS, the Pittsburgh Sleep Quality Index (PSQI) and the SF-20. In addition, participants will be instructed to maintain a glucose testing, meditation, and exercise adherence log. The glucose testing log will permit measuring consistency and adherence to treatment over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes
* Has a score above 2 on the T2D Distress Assessment Scale

Exclusion Criteria:

* Does not have type 2 diabetes
* Has a score above 2 on the T2D Distress Assessment Scale
* Cannot safely exercise
* Cannot complete the requested tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Self-Compassion | 4 weeks
  Will assess for change pre and post-intervention on standardized questionnaires on diabetes distress and self-compassion scores after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Chao, DO, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Considering sharing with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after the study, up to 1 yr after.
Access Criteria: To be determined.